CLINICAL TRIAL: NCT02910804
Title: PET-NIRF Dual Modality Imaging Guiding Surgery in Patients With Glioblastoma
Brief Title: IRDye800CW-BBN PET-NIRF Imaging Guiding Surgery in Patients With Glioblastoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Deling Li, Dr., Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BTHospital-N-005; ZIAEB000073 (NIH)
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Glioblastoma
Keywords: GBM; GRPR; IRDye800; NIRF; surgery
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-BBN-IRDye800CW PET/NIRF (Experimental): The patients were injected with 40μg/111-148 Mega-Becquerel (MBq) 68Ga-BBN-IRDye800CW in one dose intravenously and then underwent PET scan 30 min later before the operation and intraoperative 1.0 mg/ml BBN-IRDye800CW injected intravenously for near-infrared (NIR) fluorescent imaging-guided surgery.
  Interventions: Drug: 68Ga-BBN-IRDye800CW; Device: PET/NIRF; Procedure: PET/NIR fluorescent imaging-guided surgery

INTERVENTIONS:
Drug: 68Ga-BBN-IRDye800CW
  Other Names: BBN-IRDye800CW
Device: PET/NIRF
  Other Names: Positron emission tomography/Near-infrared fluorescent
Procedure: PET/NIR fluorescent imaging-guided surgery

SUMMARY:
This is an open-label positron emission tomography/near infrared (PET/NIRF) study to investigate the imaging navigation performance and evaluation efficacy of dual modality imaging probe 68Ga-BBN-IRDye800CW in glioblastoma (GBM) patients. A single dose of 40μg/111-148 Mega-Becquerel (MBq) and 1.0 mg/ml 68Ga-BBN-IRDye800CW will be injected intravenously before the operation and intraoperative respectively. Visual and semiquantitative method will be used to assess the PET images and real-time margins localization for surgical navigation.

DETAILED DESCRIPTION:
Non-invasive preoperative PET imaging evaluation and real-time fluorescence-guided surgery would be of great help in GBM patients. BBN, with the amino acid sequence of Gln-Trp-Ala-Val-Gly-His-Leu-Met-NH2, has been extensively used for the development of molecular probes for the imaging of gastrin-releasing peptide receptor (GRPR), a member of the G protein-coupled receptor family of bombesin receptors that over-expressed in various types of cancer cells including glioblastoma multiforme. For interests in clinical translation of GRPR targeting dual modality probe, an open label dual modality imaging PET/ NIFR study was designed to investigate the safety and imaging guiding performance of 68Ga-BBN-IRDye800CW in patients with GBM.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent
* MRI imaging and/or pathological evidence of Newly Diagnosed or recurrence GBM

Exclusion Criteria:

* Consisted of conditions of mental illness
* Severe liver or kidney disease with serum creatinine > 3.0 mg/dl (270 μΜ)
* Any hepatic enzyme level 5 times or more than normal upper limit
* Severe allergy or hypersensitivity to IV radiographic contrast
* Claustrophobia to accept the PET/CT scanning
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-BBN-IRDye800CW in PET imaging of GBM | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in GBM will be measured.
Margin assessment of positive tumors in NIRF fluorescent-guided surgery | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nan Ji, MD, Study Director — Beijing Tiantan Hospital, Capital Medical University Beijing 100050, China; Zhaohui Zhu, MD., Study Director — Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing 100730, China
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China